CLINICAL TRIAL: NCT00504166
Title: Alendronate Prevents Microarchitectural Deterioration of Trabecular Bone in Early Postmenopausal
Brief Title: Alendronate Prevents Microarchitectural Deterioration of Trabecular Bone in Early Postmenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: M250
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Results first posted 2011-08-10 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-07

CONDITIONS: Osteopenia; Osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Alendronate; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- alendronate sodium (Active Comparator): alendronate sodium 70 mg tablet once a week for 24 months
  Interventions: Drug: alendronate sodium
- placebo (Placebo Comparator): placebo to match alendronate sodium
  Interventions: Other: placebo comparator

INTERVENTIONS:
Drug: alendronate sodium — alendronate sodium 70 mg tablet once week for 24 months
  Other Names: fosamax
  Arms: alendronate sodium
Other: placebo comparator — placebo to match alendronate sodium one tablet once a week for 24 months
  Other Names: sugar pill
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the changes in bone structure as determined by magnetic resonance imaging measurements among early postmenopausal women after 24 months of treatment with alendronate, 70 mg once a week as compared to placebo

DETAILED DESCRIPTION:
This is a randomized, double-blind, 24-month study. Fifty-five postmenopausal women, age range of 45-65 years, with low bone density will be recruited, with half of the subjects receiving alendronate + 2800 IU of vitamin D once weekly, the other half receiving placebo + 2800 IU of vitamin D once weekly. All study subjects will receive supplemental calcium 1000 mg/day + Vitamin D 400 IU/day. Measurements of microarchitecture will be made in the wrist, ankle, and hip, and the changes in trabecular bone will be assessed at 0, 12 and 24 months. Markers of bone turnover and bone mineral density (BMD) will be used to characterize the cohort and postmenopausal changes in bone turnover and density.

ELIGIBILITY:
Inclusion Criteria:

* early postmenopausal women
* 45-65 years old
* T-score range -1.1 to -2.5 either at the lumbar spine or any hip site exclusive of Ward's triangle
* at least 3 vertebrae rom L1-L4 must be evaluable

Exclusion Criteria:

* Those at high risk for osteoporotic fracture within the next 24 months, such that randomization to a placebo would be unacceptable (e.g., prior history of hip fracture, recent symptomatic clinical vertebral fracture, or very low BMD [i.e., BMD > 2.5 SD below young normal bone mass at any site exclusive of Ward's Triangle])
* Current excessive tobacco use
* Abnormality of the esophagus which delays esophageal emptying, such as stricture or achalasia
* Gastroesophageal reflux disease sufficient to require regular medication
* Inability to stand or sit upright for at least 30 minutes once a week
* Current use of any illicit drugs or has a history of drug or alcohol abuse within the past 5 years
* Current alcohol use > 3 drinks/day
* Any of the following: hypocalcemia; severe malabsorption syndrome; moderate or severe hypertension which is uncontrolled; new onset angina or myocardial infarction within six months of entry into the study; evidence for impaired renal function defined as creatinine clearance <35 ml/min or serum creatinine greater than 1.6 mg/dL; organ transplantation; or other significant end organ diseases (genitourinary, cardiovascular, endocrine, hepatic, psychiatric, renal, hematologic, or pulmonary) which, in the opinion of the investigator, may pose an added risk to the patient or impair the patient's ability to complete the trial
* History of or evidence for metabolic bone disease (other than postmenopausal bone loss) including but not limited to vitamin D deficiency (25-hydroxy-vitamin D level <10 ng/ml), hypoparathyroidism, recent hyperthyroidism (suppressed TSH within the six months prior to entry into the study), Paget's disease of bone, Cushing's disease, osteomalacia and renal osteodystrophy
* History of cancer. However, patients with the following cancers will be considered eligible for the study: 1) superficial basal or squamous cell carcinoma of the skin which has been completely resected; 2) other malignancies completely treated without recurrence or treatment in the last 5 years, with the following exceptions: patients with a history of breast cancer (including histologic diagnosis of lobular carcinoma in situ), endometrial carcinoma, or other known or suspected estrogen-sensitive neoplasia are excluded regardless of time since treatment or disease status
* Any treatment with a bisphosphonate or parathyroid hormone; within the last 6 months: estrogen, estrogen analogues (e.g. raloxifene, tamoxifen) tibolone or anabolic steroids; Estrogen taken > 3 months ago for < 1 week is acceptable; Topical (vaginal) estrogen cream (< 2 g) used up to 2 times weekly is acceptable; Thyroid hormone, unless on a stable dose for at least six weeks before randomization with serum TSH within normal range; Fluoride treatment at a dose greater than 1 mg/day for more than 1 month at any time; given for a shorter time than one month it must have been greater than 1 year before randomization; Glucocorticoid treatment for more than one month with > 7.5 mg of oral prednisone (or the equivalent) per day within six months prior to randomization; patients who have received therapeutic glucocorticoids in the past must be considered highly unlikely to require retreatment with any dose of oral glucocorticoids for more than one month during the course of the study; Treatment with an immunosuppressant (e.g., cyclosporine, azathioprine) within the previous year.
* Current or expected treatment during the course of the study of any medication which might alter bone or calcium metabolism, including vitamin A in excess of 10,000 IU per day, or vitamin D in excess of 5,000IU per day, calcitonin, phenytoin, heparin, or lithium.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-02; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Link, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California Department of Radiology, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: Feb 2006-March 2007. Recruitment ads were posted at different UCSF campuses, senior centers, churches, train stations. We also utilized mass mailing lists, newspaper ad and radio broadcasts
Period: Overall Study
Arm/Group | Alendronate Sodium | Placebo
Started | 26 | 27
Completed | 20 | 13
Not Completed | 6 | 14
Not completed — Adverse Event | 1 | 4
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alendronate Sodium | Placebo | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 27 | 53
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 55.8 (3.9) | 55.4 (3.3) | 55.6 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 53
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 27 | 53

OUTCOME MEASURES:

1. Primary Outcome: Mean % Change From Baseline in Trabecular Number (Tb.N) by HR-pQCT
Description: Trabecular number is a three-dimensional measure of the mean inter-trabecular distance; the primary micro-architectural feature measured by high-resolution CT imaging. The parameter was calculated from scans of the distal radius and distal tibia at baseline, 12, and 24 months. The percent change from baseline over these time periods was calculated as the primary outcome measure indicating the micro-architectural status of trabecular bone.
Time Frame: Baseline, 24 months
Population: final statistical analysis was performed per protocol
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Alendronate Treatment: 70 mg of alendronate once weekly and daily 2800 IU of vitamin D3 and OSCal + D (1000 mg of calcium + 400 IU of vitamin D3)
- Placebo Treatment: daily 2800 IU of vitamin D3 and OSCal + D (1000 mg of calcium + 400 IU of vitamin D3)
Arm/Group | Alendronate Treatment | Placebo Treatment
Number analyzed (Participants) | 20 | 13
Percent change
  Distal Radius | 2.1 (7.0) | -0.6 (8.8)
  Distal Tibia | 0.9 (6.8) | 4.1 (7.5)

ADVERSE EVENTS:
Arm/Group | Alendronate Sodium | Placebo
Serious Adverse Events (participants affected / at risk) | 3/26 | 4/27
Other Adverse Events (participants affected / at risk) | 16/26 | 19/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alendronate Sodium (N=26) | Placebo (N=27)
significant bone mineral loss (Endocrine disorders) | 0 (0) | 2 (2)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anxiety attack (Psychiatric disorders) | 1 (1) | 0 (0)
Difficulty swallowing (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vitamin D overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alendronate Sodium (N=26) | Placebo (N=27)
high monocyte level (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Abnormal white cell count (Blood and lymphatic system disorders) | 5 (5) | 6 (6)
Broken tooth (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
mildly unpleasant feeling in the stomach (Gastrointestinal disorders) | 0 (0) | 1 (1)
High calcium level (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Low neutrophil count (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
High cholesterol (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
osteoarthritis of the hip (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sinus nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
sore throat (General disorders) | 0 (0) | 1 (1)
Painful urination (Renal and urinary disorders) | 0 (0) | 1 (1)
Blood-tinged urine (Renal and urinary disorders) | 0 (0) | 1 (1)
irregular heart beat (Cardiac disorders) | 0 (0) | 1 (1)
High Phosphorus level (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
vaginal odor (General disorders) | 1 (1) | 0 (0)
heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
Swelling, left ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Patches of dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
loose bowel movement (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood shot red eyes (Eye disorders) | 1 (1) | 0 (0)
swollen tongue (General disorders) | 1 (1) | 0 (0)
ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Stomach upset (Gastrointestinal disorders) | 0 (0) | 1 (1)
flu (Infections and infestations) | 0 (0) | 1 (1)
neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
dry mouth (General disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
abdominal cramping (Gastrointestinal disorders) | 1 (1) | 0 (0)
bladder infection (Renal and urinary disorders) | 0 (0) | 1 (1)
shingles, left forehead & scalp (Infections and infestations) | 1 (1) | 0 (0)
cervical vertebral disk degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Stomach flu (Gastrointestinal disorders) | 1 (1) | 0 (0)
palpitation (Cardiac disorders) | 0 (0) | 1 (1)
dental abscess (Infections and infestations) | 0 (0) | 1 (1)
Swelling, upper & lower eyelids (Eye disorders) | 0 (0) | 1 (1)
high uric acid level (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
abnormal red blood cell count (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
high alanine aminotransferase (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
high eosinophil count (Infections and infestations) | 1 (1) | 0 (0)
tooth infection #30 (Infections and infestations) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 1 (1)
cough & colds (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Low Carbon Dioxide level (General disorders) | 0 (0) | 1 (1)
High creatinine (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No